CLINICAL TRIAL: NCT03836313
Title: Does the Use of Cryoneurolysis Improve Prehabilitation Prior to Surgery Leading to Improved Postoperative Pain Management and Reduced Economic Patient Burden in Primary Total Knee Arthroplasty Patients
Brief Title: Assessing if Cryoneurolysis Improves Prehabilitation and Decreases Pain After Surgery With Less Opioid Use in TKA Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor withdrew study
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Antonia Faustina Chen, Antonia F. Chen, MD/MBA. Director of Arthroplasty Research, Principal Investigator,, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008P002629
Record Dates: First submitted 2019-02-05; First posted 2019-02-11 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Arthropathy of Knee; Pain, Joint; Arthritis Knee; Opioid Use
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- cryoneurolysis treatment (Experimental): TKA patients randomized to receive preoperative rehabilitation and cryoneurolysis treatment with the iovera° device (n=70)
  Interventions: Device: iovera°
- no cryoneurolysis treatment (standard of care) (No Intervention): TKA patients randomized to receive preoperative rehabilitation only (no cryoneurolysis treatment) (n=70)

INTERVENTIONS:
Device: iovera° — Cryoneurolysis treatment using the iovera° device targeting the anterior femoral cutaneous nerve (AFCN) and the infrapatellar branch of the saphenous nerve (ISN) will occur approximately 4 weeks before surgery by a trained member of the study staff. Treatment will occur in clinic using suggested anatomical markings to target appropriate the AFCN and infrapatellar branch of the saphenous nerve (ISN) of the operative knee.
  The iovera° device contains three 27- gauge needles, all 6.9mm in length which will indent the subjects' skin and be inserted under the subcutaneous fat about 7 mm. Lidocaine will be used for superficial anesthetic at the treatment site before the needles puncture the patient's skin.There are a total of 9 iovera° cooling cycles. Treatment will be performed unilaterally and will be guided by visualization and palpation of anatomical landmarks.
  Arms: cryoneurolysis treatment

SUMMARY:
This is a prospective, randomized control trial to evaluate the impacts of preoperative cryoneurolysis treatment on opioid consumption with prehabilitation and resulting postoperative functional improvement in patients undergoing elective primary total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Patients eligible for the study will be undergoing elective primary TKA at Brigham and Women's Hospital in Boston, MA. Study participants which meet the inclusion criteria listed above will be introduced to the study by a member of the research team in clinic when they schedule their date for surgery. If patients do not schedule an exact date for surgery at the time of their clinic visit, a member of the research team will still discuss the study with the patient so they can be called to schedule iovera° treatment once they schedule their surgical date. Patients who are interested in the study will be asked for permission to be contacted by a member of the study staff by telephone. These patients who give permission to be contacted about the study further will be called on the telephone 4-8 weeks in advance of their surgical date to assess them for their eligibility. If patients agree to participate in the study, they will be randomized to receive or not receive preoperative iovera° treatment. If the patient is eligible and agrees to participate in the study, the patient will come into clinic where informed consent will be obtained in-person at that time by a physician investigator and the patient will then receive cryoneurolysis iovera° treatment by a trained member of the study staff. Dr. Antonia Chen, Mei Xu (Dr. Chen's Physician Assistant), Dr. Wolfgang Fitz, Dr. Jeffrey Lange, Dr. Thomas Thornhill, Dr. Richard Iorio, Dr.Vivek Shah, Pierre-Emmanuel Schwab, and Brielle Antonelli will undergo an in-depth and personalized training session with a representative from Myoscience Inc. who will meet with these members in clinic in-person and review the device, the treatment procedure, and bring supplies so these specific members of the study staff can practice administering cryoneurolysis treatment before beginning the study on patients. Demographic information will be collected including the patient name, medical record number, date of birth, age, height and weight, gender, primary language, marital status, living situation, body mass index (BMI), preoperative narcotic consumption, and existing comorbidities. Randomization of patients for treatment will occur via randomized computer assignments. Patients will be randomly assigned to either the iovera° treatment group or the standard of care (SOC) group with a randomization ratio of 1:1. Patients will come in one month prior to surgery to receive prehabilitation treatment with physical therapy and undergo physical tests including quadriceps strength, timed up and go test (TUG), single leg stance, balance, and timed horizontal leg hold (quadriceps endurance test). Patients will also fill-out patient reported outcome measures (PROMs), such as KOOS, PROMIS 10, visual analog scale (VAS), the Pain Catastrophizing Scale (PCS), and EQ-5D. The first functional test and completion of PROMs will occur before iovera° treatment takes place at the first visit when subjects come into the clinic to receive iovera° treatment. The second functional test and completion of PROMs will occur on subject's day of surgery before the procedure, and the third set of functional test and completion of PROMs will be postoperatively at the subject's follow-up visit in clinic between 2-6 weeks.

The iovera° device is FDA approved (510(k) [#K142866]) for treatment of peripheral nerves for pain and for treatment of the pain and symptoms of knee osteoarthritis for up to 90 days (K161835). This device will be used according to its FDA labeling in patients with pain - hence why they are having a knee replacement, which would be pain due to osteoarthritis.

Cryoneurolysis treatment using the iovera° device targeting the anterior femoral cutaneous nerve (AFCN) and the infrapatellar branch of the saphenous nerve (ISN) will occur approximately 4 weeks before surgery by a trained member of the study staff (as mentioned above). Treatment will occur in the clinic setting using suggested anatomical markings to target appropriate the AFCN and infrapatellar branch of the saphenous nerve (ISN) of the operative knee. Patients are not sedated and will be asked to identify the painful locations with one finger which will be marked. The study staff member administering treatment will push on these locations to confirm that the marked areas are where the patient experiences pain and responds regarding their sensation and cessation of the pain signaling. This will confirm the correct location for the investigators which will also be confirmed with the aforementioned anatomical locations of the appropriate nerve branches.

The iovera° device contains three 27- gauge needles, all 6.9mm in length which will indent the subjects' skin and be inserted under the subcutaneous fat about 7 mm. Other tissues which may be impacted in addition to the subcutaneous fat are the dermis and epidermis. Muscle is rarely involved. Given that the needles are only 6.9mm in length, there is minimal possibility of reaching and affecting fascia, muscle, or vascular structures in the area which will be treated. All of these tissues impacted, subcutaneous fat are the dermis and epidermis, recover or are unaffected by the cooling based on the safety profile of safety profile of cryoanalgesia. Some patients who may have variations in anatomy, particularly in thickness of subcutaneous fat, will undergo the same procedure, but the investigator will push the handpiece down to displace the subcutaneous fat. Furthermore, surgeons in this practice exercise a patient BMI cut off of 40 kg/m2, which will minimize the amount of subcutaneous fat. Lidocaine will be used for superficial anesthetic at the treatment site before the needled puncture the patient's skin and no additional nerve block will be used at this time. Each subject will undergo a total of 9 treatments, or cooling cycles, using the iovera° device since each nerve branch has 2-3 sites per branch due to the anatomy of these nerve branches determined using determined anatomical markings. Treatment will be performed unilaterally and will be guided by visualization and palpation of anatomical landmarks. With there being 3 nerve branches with about 3 treatment sites per branch, the total number of treatments per subject is 9 with each treatment lasting about 1 minute, totaling 9-10 minutes of active treatment. The amount of time estimated for the entire treatment is 20 minutes. Investigators will know that they are hitting the targeted nerve since the subject is not sedated and can report a parasthesia response in real-time when the nerve is frozen.

Surgical data including date of surgery, laterality, anesthesia type, pericapsular injections, tourniquet (yes/no), morphine equivalents used in hospital, and discharge location will be collected for each participant. All other standard of care FDA approved medications and nerve blocks will be used in the operating room and postoperatively as needed depending upon the need of each individual patient as determined by the surgeon. These medications and nerve blocks commonly include bupivacaine, ropivacaine, toradol, clonidine, epinephrine, meloxicam, tylenol, oxycodone, vicodin, percocet, tramadol, toradol, dilaudid, morphine, lyrica, celebrex, and gabapentin.

All participants will receive a standard 7 days of opioid medication with 40 pills after surgery. Subjects will be instructed to take their prescribed pain medication (Oxycodone 5-10mg or dilaudid 1-2mg) every 4-6 hours as need. Surveys distributed through RedCap will be sent to each patient daily via email to track and monitor opioid consumption and physical therapy sessions daily, once a day preoperatively with 7 short questions for approximately 4 weeks (from their iovera° treatment until their scheduled date of surgery), and once a day postoperatively with 10 short questions for 6 weeks for a total of 70 surveys per patient for the entire study. Each survey should take no longer than a few minutes to complete. Follow-up visits will take place at 2-6 weeks after surgery for every participant, with one more survey follow-up at 12 weeks. At each follow-up visit, participants will undergo the same preoperative physical tests and fill-out each PROM. The postoperative data that will be collected will consist of physical therapy utilized, narcotic consumption (morphine equivalents), if patients used opioid medication 60 days prior to surgery or not, time to return to activities of daily living, time off of assistive walking devices, and 90-day complications (readmission, reoperation, emergency room visits) which will determine estimated financial costs of both treatment groups. The investigators will follow patients postoperatively to evaluate their pain scores to determine if there are differences in pain scores between the SOC group and the iovera° group and to specifically see if there is increased pain in the iovera° group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age >= 18 years of age and undergoing elective unilateral primary total knee arthroplasty
* All subjects who are willing to comply with the requirements of the study and provide informed consent prior to enrollment. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study must be obtained before data collection.

Exclusion Criteria:

* Subjects that are undergoing bilateral TKA or revision TKA
* Pregnant women and vulnerable individuals.
* Patients who cannot undergo cryoneurolysis (i.e. Patients with cryoglobulinemia, paroxysmal cold hemoglobinuria, cold urticaria, Raynaud's disease, open/ infected wounds at or near the treatment site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
narcotic consumption after surgery | 4 weeks
  determine if preoperative iovera° cryoneurolysis treatment with prehabilitation decreases opioid medication consumption based on morphine equivalents consumed within the first 4 weeks after surgery

SECONDARY OUTCOMES:
knee pain after surgery: Visual Analogue Scale (VAS) for pain | 3 months
  Determine if preoperative iovera° cryoneurolysis treatment with prehabilitation decreases knee pain based on the VAS pain scale 3 months after surgery. The VAS is used to assess the intensity and frequency of pain. The scale is a line of 10cm and the distance of the line which lines up with the patient's reported pain is measured in millimeters. The scale is interpreted as follows: no pain (0-4mm), mild pain (5-44mm), moderate pain (45-74mm), and severe pain (75-100mm).
patient quadriceps strength | 3 months
  Determine if preoperative iovera° cryoneurolysis treatment with prehabilitation increases patient quadriceps strength as determined by the muscle strength scale (0-5), with 0 being no strength and 5 being more strength,comparing preoperative strength, to strength at the time of surgery and 3 months postoperatively
postoperative pain (measured by the Knee Injury and Osteoarthritis Outcome Score (KOOS)). | 3 months
  Determine if preoperative iovera° cryoneurolysis treatment with prehabilitation improves postoperative pain compared to patients who do not undergo treatment based on patient reported outcome scores using KOOS at 3 months postoperatively. KOOS assesses short and long term patient satisfaction and pain after knee injury/ surgery associated with primary osteoarthritis. KOOS is scored using 5 subscales (pain, symptoms, activities of daily living, sport / recreational activity, and quality of life. Each subcategory is scored from 0 (no problems) to 4 (extreme problems). Those scores are determined as the sum of included items per subcomponent. These scores are converted to a 0-100 scale with 0 being extreme problems and 100 representing no knee problems.
patient discharge location after surgery (home versus rehabilitation or skilled nursing facilities) | 3 months
  Evaluate if preoperative treatment with iovera° affects discharge location (home versus rehabilitation or skilled nursing facilities) between patients who do and do not undergo iovera° cryoneurolysis treatment
general health and physical function (measured by Patient- Completed Health Outcomes Measurement Information System (PROMIS-10)) | 3 months
  Determine if preoperative iovera° cryoneurolysis treatment with prehabilitation improves postoperative general health and physical function compared to patients who do not undergo treatment based on patient reported outcome scores using PROMIS-10 at 3 months postoperatively. PROMIS-10 assesses overall general health, including physical, mental, and social health along with pain, fatigue, and patient-reported quality of life. This scale has 10 items which are each scored separately and represented with 5 points. The scores are then grouped into 2 domains - Global Physical Health Score and Global Mental Health Score. A T-score is used to standardize these scores to the general population where higher scores represent healthier patients. The average score for the U.S. population is 50.
patient physical therapy use after surgery | 3 months
  Evaluate if preoperative treatment with iovera° affects use of physical therapy after surgery in terms of number of patient physical therapy visits determined by a daily electronic custom-made emailed questionnaire in patients who do and do not undergo iovera° cryoneurolysis treatment in the postoperative period 3 months after surgery. The questionnaire will ask patients if they went to physical therapy on a daily basis and if they completed their exercises. This is not a scale. We are recording the number of physical therapy sessions that a patient engages in postoperatively, without a limit.

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Chen, MD/MBA, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No
There will no IPD data shared, and only aggregated data will be used.

REFERENCES:
- [Result] Dasa V, Lensing G, Parsons M, Harris J, Volaufova J, Bliss R. Percutaneous freezing of sensory nerves prior to total knee arthroplasty. Knee. 2016 Jun;23(3):523-8. doi: 10.1016/j.knee.2016.01.011. Epub 2016 Feb 10. PMID 26875052
- [Result] Barnard D. The effects of extreme cold on sensory nerves. Ann R Coll Surg Engl. 1980 May;62(3):180-7. PMID 7396346
- [Result] Gabriel RA, Finneran JJ, Asokan D, Trescot AM, Sandhu NS, Ilfeld BM. Ultrasound-Guided Percutaneous Cryoneurolysis for Acute Pain Management: A Case Report. A A Case Rep. 2017 Sep 1;9(5):129-132. doi: 10.1213/XAA.0000000000000546. PMID 28509777
- [Result] Ilfeld BM, Gabriel RA, Trescot AM. Ultrasound-guided percutaneous cryoneurolysis providing postoperative analgesia lasting many weeks following a single administration: a replacement for continuous peripheral nerve blocks?: a case report. Korean J Anesthesiol. 2017 Oct;70(5):567-570. doi: 10.4097/kjae.2017.70.5.567. Epub 2017 Feb 3. PMID 29046778
- [Result] Ilfeld BM, Preciado J, Trescot AM. Novel cryoneurolysis device for the treatment of sensory and motor peripheral nerves. Expert Rev Med Devices. 2016 Aug;13(8):713-25. doi: 10.1080/17434440.2016.1204229. Epub 2016 Jul 13. PMID 27333989
- [Result] Inacio MCS, Paxton EW, Graves SE, Namba RS, Nemes S. Projected increase in total knee arthroplasty in the United States - an alternative projection model. Osteoarthritis Cartilage. 2017 Nov;25(11):1797-1803. doi: 10.1016/j.joca.2017.07.022. Epub 2017 Aug 8. PMID 28801208
- [Result] Pua YH, Ong PH. Association of early ambulation with length of stay and costs in total knee arthroplasty: retrospective cohort study. Am J Phys Med Rehabil. 2014 Nov;93(11):962-70. doi: 10.1097/PHM.0000000000000116. PMID 24879549
- [Result] Radnovich R, Scott D, Patel AT, Olson R, Dasa V, Segal N, Lane NE, Shrock K, Naranjo J, Darr K, Surowitz R, Choo J, Valadie A, Harrell R, Wei N, Metyas S. Cryoneurolysis to treat the pain and symptoms of knee osteoarthritis: a multicenter, randomized, double-blind, sham-controlled trial. Osteoarthritis Cartilage. 2017 Aug;25(8):1247-1256. doi: 10.1016/j.joca.2017.03.006. Epub 2017 Mar 20. PMID 28336454
- [Result] Trescot AM. Cryoanalgesia in interventional pain management. Pain Physician. 2003 Jul;6(3):345-60. PMID 16880882
- [Result] Zhou L, Kambin P, Casey KF, Bonner FJ, O'Brien E, Shao Z, Ou S. Mechanism research of cryoanalgesia. Neurol Res. 1995 Aug;17(4):307-11. doi: 10.1080/01616412.1995.11740333. PMID 7477749
- [Result] Zhou L, Shao Z, Ou S. Cryoanalgesia: electrophysiology at different temperatures. Cryobiology. 2003 Feb;46(1):26-32. doi: 10.1016/s0011-2240(02)00160-8. PMID 12623025